CLINICAL TRIAL: NCT05598697
Title: Economic Evaluation of the Men Engagement in Women Empowerment (MEWE) Intervention (MEWE-EE)
Brief Title: Economic Evaluation of the MEWE Intervention
Acronym: MEWE-EE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Economics and Political Science (Other)
Collaborators: Aga Khan University (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Giulia Ferrari, Assistant Professorial Research Fellow, London School of Economics and Political Science
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 108137
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Depression; Mental Health Issue; Intimate Partner Violence; Domestic Violence; Gender-based Violence; Rape Sexual Assault; Battered Women
Keywords: violence; abuse; coercion; assault; aggression; gender; women; girl; wife; partner; spouse; sexual; physical; psychological; economic
MeSH Terms: conditions — Depression; Aggression; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cash Transfers only (Active Comparator): Participants allocated to this arm receive cash transfers. They are clients of a nation-wide cash transfer program.
  Interventions: Other: Cash transfer to adult females
- Cash Transfers + LSB curriculum for females clients only (Experimental): Participants allocated to this arm receive cash transfers and access to LSB curriculum training. Female cash transfer recipients attend 10 life-skills building sessions. Sessions are held weekly and are 90 minutes long. Two trained facilitators run the session for groups of 10 women over a ten-week period.
  Interventions: Behavioral: Life Skills Building (LSB) curriculum for females; Other: Cash transfer to adult females
- Cash Transfers + LSB curriculum for females clients and their husbands (Experimental): Participants allocated to this arm receive cash transfers and access to LSB curriculum training in gender-segregated groups. Men and women attend 10 life-skills building sessions in parallel. Sessions are held weekly and are 90 minutes long. Two trained facilitators, whose gender matches the participants', run the session for groups of 10 women or men over a ten-week period.
  Interventions: Behavioral: Life Skills Building (LSB) curriculum for males; Behavioral: Life Skills Building (LSB) curriculum for females; Other: Cash transfer to adult females

INTERVENTIONS:
Behavioral: Life Skills Building (LSB) curriculum for males — The LSB curriculum offers ten weekly 90-minute sessions. Topics include effective communication, gender roles, power dynamics in the household; work-life balance and time management; conflict resolution; household decision making. The LSB teachers are trained in facilitation techniques to deliver the sessions.
  All male study participants attending LSB curriculum classes are married to BISP-CT clients.
  For men, the MEWE intervention provides access to the LSB curriculum only.
  Other Names: MEWE males
  Arms: Cash Transfers + LSB curriculum for females clients and their husbands
Behavioral: Life Skills Building (LSB) curriculum for females — The LSB curriculum offers ten weekly 90-minute sessions. Topics include effective communication, gender roles, power dynamics in the household; work-life balance and time management; conflict resolution; household decision making. The LSB teachers are trained in facilitation techniques to deliver the sessions.
  All female study participants attending LSB curriculum classes are BISP-CT clients.
  For females, the MEWE intervention comprises access to LSB curriculum + BISP CTs.
  Other Names: MEWE females
  Arms: Cash Transfers + LSB curriculum for females clients and their husbands; Cash Transfers + LSB curriculum for females clients only
Other: Cash transfer to adult females — The BISP intervention offers access to quarterly unconditional cash transfers to adult females.
  Other Names: BISP-CT

SUMMARY:
Cash transfers have shown promise in preventing intimate partner violence, and in reducing recipients' stress levels. Cash transfers with behavioral or psychological interventions have shown limited effectiveness at reducing stress in some African countries. Little is known of the cost-effectiveness of interventions delivered alongside cash transfer programs. The MEWE economic evaluation sub-study (MEWE-EE) runs alongside MEWE, a three-arm cluster-randomized controlled trial in Sindh, Pakistan. MEWE-EE will assess the costs and cost-effectiveness of delivering a cash-transfer program (BISP-CT) combined with a life-skills building curriculum (LSB curriculum), compared to the BISP-CT alone. The LSB curriculum is offered to either women who receive BISP-CT, or to women who receive BISP-CT and their husbands.

ELIGIBILITY:
Inclusion Criteria:

* In receipt of Benazir Income Support Program (BISP) cash transfers (CTs)
* Parity: have at least one child, at least 18 months old

Exclusion Criteria:

* Plan for the family to migrate out of the village within the next 2 years

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1536 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Incremental cost incurred per disability adjusted life year (DALY) averted: provider perspective | 12 months post randomisation
  Incremental cost per disability-adjusted life year (DALY) averted by the intervention compared to the control group from a provider perspective at 12 months from baseline. DALYs and costs will also be modelled up to a ten-year horizon using a Markov model.
Incremental cost incurred per disability adjusted life year (DALY) averted: societal perspective | 12 months post randomisation
  Incremental cost per disability-adjusted life year (DALY) averted by the intervention compared to the control group from a societal perspective at 12 months from baseline. DALYs and costs will also be modelled up to a ten-year horizon using a Markov model.

SECONDARY OUTCOMES:
Mean cost of intervention delivery | 12 months post randomisation
  Cost of intervention delivery for different intervention models per patient, by category, annuitised
Mean cost of LSB session | 12 months post randomisation
  Average cost of LSB session delivery for different intervention models, annuitised
Total incremental cost of the intervention in a research setting | 12 months post randomisation
  Total additional cost of the intervention compared to the BISP-CT only for the study population and by intervention type during the research period.
Total incremental cost of the intervention in the modelling cohort | 12 months post randomisation
  Total additional cost of the intervention for the modelling cohort by intervention type over a ten-year period.
Incremental cost incurred per disability adjusted life year (DALY) averted at scale: provider perspective | 12 months post randomisation
  Incremental cost per disability-adjusted life year (DALY) averted by the intervention compared to the control group from a provider perspective at scale.
Incremental cost incurred per disability adjusted life year (DALY) averted at scale: societal perspective | 12 months post randomisation
  Incremental cost per disability-adjusted life year (DALY) averted by the intervention compared to the control group from a societal perspective at scale.

CONTACTS AND LOCATIONS:
Overall Officials: Giulia Ferrari, PhD, Principal Investigator — London School of Economics & Political Science
Locations (1):
- Mirpur Sakro, Thatta, Sindh, Pakistan